CLINICAL TRIAL: NCT04268693
Title: Bisphenol and Phthalate Exposures in Women With Triple Negative Breast Cancer Receiving Doxorubicin Chemotherapy - a Pilot Study
Brief Title: Bisphenol and Phthalate Exposures in Triple Negative Breast Cancer
Acronym: EDC-TNBC
Status: Withdrawn | Type: Observational
Why Stopped: Study never initiated due to COVID pandemic, staffing changes
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Kimberly Robien, Associate Professor, George Washington University
Other Study IDs: NCR191600
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Triple Negative Breast Cancer
Keywords: bisphenol; phthalate; doxorubicin
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: urinary bisphenol and phthalate levels
  Interventions: Other: urine collection

INTERVENTIONS:
Other: urine collection — Collect three urine samples either in the clinic or at home. This will occur prior to starting neoadjuvant chemotherapy, and again at the end of the scheduled course of neoadjuvant chemotherapy.

SUMMARY:
In this observational pilot study urine samples will be collected from women receiving neoadjuvant chemotherapy with doxorubicin for triple negative breast cancer to determine whether: 1) exposures bisphenol and phthalate levels change over the course of neoadjuvant chemotherapy, and 2) levels differ between black women and those of other racial groups.

The hypothesis is that bisphenol and phthalate levels will be similar to those of the general US female population at the time of diagnosis, however levels will increase during treatment due to exposure to plastics in the medical setting. The investigators also hypothesize that because of differences in personal care product use, black women may have higher urinary levels of bisphenols and phthalates prior to starting chemotherapy.

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC) is an aggressive breast cancer subtype that does not express estrogen, progesterone, or the human epidermal growth factor (HER2/neu) receptors, and has a low overall survival rate compared to other types of breast cancer.

Unlike hormone and HER2/neu positive breast cancers, targeted therapies are not available for TNBC. Thus, the systemic chemotherapeutic agent doxorubicin is widely used for the treatment of TNBC. However, doxorubicin resistance is common, and leads to poorer treatment outcomes.

Understanding factors that contribute to doxorubicin resistance is critical to improving cancer treatment outcomes among women with TNBC. Pre-clinical in vitro studies indicate that exposure to endocrine disrupting chemicals, such as bisphenols and phthalates, contribute to doxorubicin resistance, but these findings have not been evaluated in humans.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stage I - III triple negative breast cancer
* scheduled to receive a neoadjuvant chemotherapy regimen including doxorubicin
* receiving treatment at the George Washington University Cancer Center

Exclusion Criteria:

* diagnosis of other types of breast cancer
* not scheduled to receive doxorubicin as part of the neoadjuvant chemotherapy regimen
* not planning to receive neoadjuvant chemotherapy at the George Washington University Cancer Center

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women being treated at the George Washington University for stage I - III triple negative breast cancer who are scheduled to receive a neoadjuvant chemotherapy regimen containing doxorubicin.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
urinary bisphenol and phthalate metabolite levels | baseline
  quantification of bisphenol and phthalate metabolites by liquid chromotography-tandem mass spectrometry
urinary bisphenol and phthalate metabolite levels | post-neoadjuvant chemotherapy (either 16 or 20 weeks)
  quantification of bisphenol and phthalate metabolites by liquid chromotography-tandem mass spectrometry
change from baseline urinary bisphenol and phthalate levels at end of neoadjuvant chemotherapy | baseline and post-neoadjuvant chemotherapy (16 or 20 weeks)
  percent of change in urinary bisphenol and phthalate levels from pre- to post-neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Kim Robien, PhD, RD, Principal Investigator — Milken Institute School of Public Health, George Washington University
Locations (1):
- Milken Institute School of Public Health, George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Will not share data until study is complete and all data deidentified